CLINICAL TRIAL: NCT00686504
Title: An Open Label, Non-randomized Positron Emission Tomography (PET) Study With [11C]AZ12713580 to Determine Central mGluR5 Receptor Occupancy of AZD2066 After Oral Administration to Healthy Subjects
Brief Title: Positron Emission Tomography (PET) Study With [11C]AZ12713580 to Determine Central mGluR5 Receptor Occupancy of AZD2066
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director, Emerging Analgesia, AstraZeneca R&D Södertälje, Sweden
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0475C00013; EudractCT 2008-000064-17
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Pain; PET; Phase 1; Analgesia; Positron Emission Tomography; mGlu5 receptor; Dose finding; Analgesia/Pain
MeSH Terms: conditions — Pain; Agnosia | interventions — AZD2066

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD2066 — single dose of oral dose, 3 times per subject
Drug: radioligand [11C] AZ12713580 — single dose of iv administered 4 times per subject (3 times together with AZD2066)

SUMMARY:
The study is carried out in order to determine the relationship between AZD2066 exposure and mGluR5 receptor occupancy in the brain and to demonstrate that AZD2066 can displace [11C]AZ12713580 from mGluR5 binding-sites in the Central Nervous System

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* BMI (Body Mass Index) of ≥19 to ≤28 kg/m2 and weight of ≥50 to ≤100 kg
* Normal MRI (Magnetic Resonance Imaging) scan at visit 2

Exclusion Criteria:

* History of previous or ongoing psychiatric disease or condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders
* History of psychotic disorder among first degree relatives (parents, siblings)
* History of use of antipsychotic, antidepressant or anxiolytic (anxiety treatment) drugs, prescribed or non-prescribed use. History of antidepressants or anxiolytics for non-psychiatric conditions such as pain or post-operative insomnia is allowed

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography using the radioligand radioligand [11C]AZ12713580 | 4 times

SECONDARY OUTCOMES:
To investigate the safety and tolerability of AZD2066 by assessment of Adverse Events (AEs), vital signs measurements (blood pressure and pulse), electrocardiogram (ECG), physical examination, clinical chemistry, haematology and urinalysis. | 7 visits with tests for all subjects. Some tests will be done several times per visit. All tests will not be performed at every visit.
To investigate pharmacokinetics of AZD2066 | 15 times per subject. Up to 48 hours each time

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, Principal Investigator — Astrazeneca Clinical Pharmacology Unit, Stockholm, Sweden; Sophia Bengtsson, Study Director — AstraZeneca R&D, Study Delivery, Clinical Development, Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden